CLINICAL TRIAL: NCT03313089
Title: Nutritional Impact of a Project on Food Security and Nutrition in Children of 6 Months to 5 Years of Age Receiving Home Fortification With Micronutrient Powders in Nariño, Colombia
Brief Title: Nutritional Impact of a Project on Food Security and Nutrition in Children Receiving Micronutrient Powders in Colombia
Status: Completed | Type: Observational
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: International Development Research Centre, Canada (Other Government); McGill University (Other)
Responsible Party: Principal Investigator, Nathalie Ospina, Master Student, Universidad Nacional de Colombia
Other Study IDs: 37460
Record Dates: First submitted 2017-10-09; First posted 2017-10-18 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Hemoglobin; Anemia
Keywords: micronutrient powders; spinkles; nutrition; food security program; nutritional program; hemoglobin; anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PSAN + MNP: PSAN ("Papas más nutritivas" project) + MNP (micronutrients powders):
  Children of the families beneficiaries of Community Schools of Family Agriculture of the municipalities of Cumbal, Carlosama Guachucal and Túquerres, who are part of the project "Papas más nutritivas" and exposed to project activities in which they work on topics related to food and nutritional security, equity and gender, production and entrepreneurship, Additionally, the home fortification with MNP that is 12 months in total approximately, will be made 2 deliveries of 60 doses (specified in the "MNP only" group). After the delivery of MNP, advising, measurements of weight and height, clarification of doubts regarding fortification with MNP, nutrition education, and accompaniment by the project staff will take place.
  Interventions: Behavioral: "Papas más nutritivas" (PSAN)
- MNP only: Cohort of exposed to MNP (micronutrients powders):
  Children who will receive MNP delivered through the hospital or institutional health service providers of the municipalities of Guachucal and Carlosama, following the protocol for the home fortification with MNP that is 12 months in total approximately, will be made 2 deliveries of 60 doses: the first period consists of the taking of MNP for 2 months, followed by a rest period of 4 months and continues again by another MNP intake for 2 months and rest for 4 months, and exposed to dissemination of basic information with regard to MNP and monitoring by growth and development that is routinely performed by health staff.

INTERVENTIONS:
Behavioral: "Papas más nutritivas" (PSAN) — Activities of the project "Papas más nutritivas"
  Groups: PSAN + MNP

SUMMARY:
The effectiveness of micronutrient powders or MNP as a strategy for the prevention of micronutrient deficiencies has been described in the literature. However, few studies have shown the impact of the inclusion of other simultaneous actions on the different dimensions of food and nutritional security (as in the case of the project "Papas más nutritivas") that will contribute to the improvement of nutritional status, obtaining potentially greater benefits.

The objective is to establish the existence of difference in hemoglobin values (and other biochemical parameters as secondary outcomes) among children aged 6 months to 5 years who receive home fortification with micronutrient powders (MNP) belonging to the project "Papas más nutritivas", and children with home fortification with MNP but not belonging to the project.

DETAILED DESCRIPTION:
Micronutrient deficiency is a public health problem. At the national level according to ENSIN 2010, in Colombia the prevalence of anemia in children of 6 to 59 months is 27.5%; of 24.3% for vitamin A deficiency in children between 1 and 4 years of age; and in the case of zinc deficiency, the prevalence is of 43.3% of children under 5 years of age. According to FAO and WHO, different strategies for overcoming micronutrient deficiencies need to be combined and balanced in order to achieve maximum impact.

The project "Papas más nutritivas" ("Ampliación de la producción de papas amarillas más nutritivas en Colombia (CIFSRF phase 2) / Scaling up synergetic strategies in agriculture and nutrition in rural communities of Colombia") funded by the IDRC-International Development Research Center, through the Canadian International Food Security Research Fund (CISFR) and implemented by the McGILL University Canada and the Universidad Nacional de Colombia involve, in addition to the expansion of production of the new varieties of yellow potatoes, other activities such as Community Schools of Family Agriculture, training schools of leader and managers in sovereignty and food and nutritional security, strengthening of the shagra (home garden) and home fortification with micronutrients powders, seeking to improve the quality of life and nutritional status of families of potato producers for the scope of the food and nutritional security.

The effectiveness of micronutrient powders or MNP as a strategy for the prevention of micronutrient deficiencies has been described in the literature. However, few studies have shown the impact of the inclusion of other simultaneous actions on the different dimensions of food and nutritional security (as in the case of the project "Papas más nutritivas") that will contribute to the improvement of nutritional status, obtaining potentially greater benefits.

Objective: To establish the existence of difference in hemoglobin values among children aged 6 months to 5 years who receive home fortification with micronutrient powders (MNP) belonging to the project "Papas más nutritivas", and children with home fortification with MNP but not belonging to the project.

Methodology: Prospective cohort. Two groups are established: the first, children exposed to the activities of the project "Papas más nutritivas" + MNP (PSAN+MNP group) , and the second, children exposed only to MNP (MNP group). We will try to include 140 children (70 for each of the groups), this sample gives us a power of 90% to find a delta of 0.5.

Blood samples will be obtained to evaluate the biochemical parameters: Hemoglobin (determined by HemoCue), Ferritin, Transferrin, Zinc, vitamin A, C-reactive-ultrasensitive protein, before MNP fortification and when it finished.

For statistical analysis, a descriptive analysis of both PSAN + MNP and MNP groups will be carried out on sociodemographic variables, health status and nutritional status. The continuous variables will be expressed with their measures of central tendency and dispersion, for the categorical variables absolute and relative frequencies will be used. The hypothesis of equality of pre and post treatment hemoglobin differences between the groups (PSAN + MNP versus MNP) will be analyzed using a Student t test or Mann Whitney test, depending on whether the data follow a normal distribution. A statistically significant p value corresponding to 0.05 will be considered. The other secondary outcome variables (vitamin A, zinc, ferritin, transferrin) will be similarly analyzed. In order to control the systematic differences in the baseline characteristics between the intervention and control groups, it is proposed to use Propensity Score, which will include the variables of sex, age and other sociodemographic and nutritional variables considered potentially confusing. The score of the propensity score model will be used as a covariate in a linear regression model where it will be adjusted further by the pre-test values of the intervention (ANCOVA). An unadjusted preliminary analysis (initially described) will be presented and then a new analysis with the proposed adjustment. An additional analysis will be performed for the ferritin variable excluding patients with high CRP values.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls of 6 months to 5 years of age receiving home fortification with micronutrient powders.

Exclusion Criteria:

* Children who are consuming nutritional complements or supplements.
* Children undergoing treatment for anemia or other micronutrient deficiencies.

Ages: 6 Months to 5 Years | Sex: All
Age Groups: Child
Study Population: Boys and girls of 6 months to 5 years of age inhabitants of municipalities: Carlosama, Guachucal, Túquerres and Cumbal in the department of Nariño,
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2017-11-26 (Actual); Study Completion 2017-11-26 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin concentration | Baseline and after 12 months approximately
  g/dL

SECONDARY OUTCOMES:
Vitamin A (change in serum retinol concentration) | Baseline and after 12 months approximately
  μg / dL
Change in zinc concentration | Baseline and after 12 months approximately
  μg / dL
Change in transferrin concentration | Baseline and after 12 months approximately
  mg / dL
Change in ferritin concentration | Baseline and after 12 months approximately
  μg / L

CONTACTS AND LOCATIONS:
Overall Officials: Sara E. Del Castillo Matamoros, Professor, Study Director — Universidad Nacional de Colombia; Javier H. Eslava Schmalbach, Professor, Study Director — Universidad Nacional de Colombia; Nathalie Ospina Lizarazo, Student, Principal Investigator — Universidad Nacional de Colombia
Locations (1):
- Universidad Nacional de Colombia, Bogotá, Colombia

REFERENCES:
- [Background] Ministerio De Salud y Protección Social. Estrategia Nacional para la Prevención y Control de las Deficiencias de Micronutrientes en Colombia 2014 - 2021. Bogotá D.C., Colombia. 2015.
- [Background] World Health Organization and Food and Agriculture Organization of the United Nations. Guidelines on Food Fortification with Micronutrients. Editado por Lindsay Allen y cols.
- [Background] Black R. Micronutrient deficiency--an underlying cause of morbidity and mortality. Bull World Health Organ. 2003;81(2):79. Epub 2003 Mar 25. No abstract available. PMID 12751414
- [Background] Ministerio de la Protección Social. Instituto Colombiano de Bienestar Familiar. ENSIN 2010- Encuesta Nacional de Situación Nutricional en Colombia 2010. Ed. Bogotá: 2011.
- [Background] OMS. Directriz: Uso de micronutrientes en polvo para la fortificación domiciliaria de los alimentos consumidos por lactantes y niños de 6 a 23 meses de edad. Ginebra, Organización Mundial de la Salud, 2012.
- [Background] Zlotkin SH, Schauer C, Christofides A, Sharieff W, Tondeur MC, Hyder SM. Micronutrient sprinkles to control childhood anaemia. PLoS Med. 2005 Jan;2(1):e1. doi: 10.1371/journal.pmed.0020001. PMID 15696200
- [Background] De-Regil LM, Suchdev PS, Vist GE, Walleser S, Pena-Rosas JP. Home fortification of foods with multiple micronutrient powders for health and nutrition in children under two years of age. Cochrane Database Syst Rev. 2011 Sep 7;(9):CD008959. doi: 10.1002/14651858.CD008959.pub2. PMID 21901727
- [Background] Hotz C, Pelto G, Armar-Klemesu M, Ferguson EF, Chege P, Musinguzi E. Constraints and opportunities for implementing nutrition-specific, agricultural and market-based approaches to improve nutrient intake adequacy among infants and young children in two regions of rural Kenya. Matern Child Nutr. 2015 Dec;11 Suppl 3(Suppl 3):39-54. doi: 10.1111/mcn.12245. PMID 26778801
- [Background] Inayati DA, Scherbaum V, Purwestri RC, Wirawan NN, Suryantan J, Hartono S, Bloem MA, Pangaribuan RV, Biesalski HK, Hoffmann V, Bellows AC. Combined intensive nutrition education and micronutrient powder supplementation improved nutritional status of mildly wasted children on Nias Island, Indonesia. Asia Pac J Clin Nutr. 2012;21(3):361-73. PMID 22705425
- [Background] Attanasio OP, Fernandez C, Fitzsimons EO, Grantham-McGregor SM, Meghir C, Rubio-Codina M. Using the infrastructure of a conditional cash transfer program to deliver a scalable integrated early child development program in Colombia: cluster randomized controlled trial. BMJ. 2014 Sep 29;349:g5785. doi: 10.1136/bmj.g5785. PMID 25266222
- [Background] Andrew A, Attanasio O, Fitzsimons E, Rubio-Codina M. Why is multiple micronutrient powder ineffective at reducing anaemia among 12-24 month olds in Colombia? Evidence from a randomised controlled trial. SSM Popul Health. 2016 Mar 7;2:95-104. doi: 10.1016/j.ssmph.2016.02.004. eCollection 2016 Dec. PMID 29349132
- [Background] Jack SJ, Ou K, Chea M, Chhin L, Devenish R, Dunbar M, Eang C, Hou K, Ly S, Khin M, Prak S, Reach R, Talukder A, Tokmoh LO, Leon de la Barra S, Hill PC, Herbison P, Gibson RS. Effect of micronutrient sprinkles on reducing anemia: a cluster-randomized effectiveness trial. Arch Pediatr Adolesc Med. 2012 Sep;166(9):842-50. doi: 10.1001/archpediatrics.2012.1003. PMID 22801933
- [Background] Aboud FE, Akhter S. A cluster-randomized evaluation of a responsive stimulation and feeding intervention in bangladesh. Pediatrics. 2011 May;127(5):e1191-7. doi: 10.1542/peds.2010-2160. Epub 2011 Apr 18. PMID 21502222
- [Background] Avula R, Frongillo EA, Arabi M, Sharma S, Schultink W. Enhancements to nutrition program in Indian integrated child development services increased growth and energy intake of children. J Nutr. 2011 Apr 1;141(4):680-4. doi: 10.3945/jn.109.116954. Epub 2011 Feb 23. PMID 21346106
- [Background] Osei AK, Pandey P, Spiro D, Adhikari D, Haselow N, De Morais C, Davis D. Adding multiple micronutrient powders to a homestead food production programme yields marginally significant benefit on anaemia reduction among young children in Nepal. Matern Child Nutr. 2015 Dec;11 Suppl 4(Suppl 4):188-202. doi: 10.1111/mcn.12173. PMID 25682798
- [Background] Del Castillo SE, Mosquera T, Suárez EL, Heredia P. Nutritional Situation of Rural Communities in Nariño, Colombia 2013. Food and Nutrition Sciences (5): 1521-1528, 2014
- See also: Sitio Web. Proyecto Seguridad Alimentaria Nutricional S.A.N. Nariño. — http://www.seguridadalimentarianarino.unal.edu.co